CLINICAL TRIAL: NCT02668003
Title: The MAintaining MusculOskeleTal Health (MAmMOTH) Study
Brief Title: The Maintaining Musculoskeletal Health Study
Acronym: MAmMOTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 02/004/14; 20748 (Other Grant/Funding Number: Arthritis Research UK); 16/SW/0019 (Other: National Research Ethics Service); 184303 (Other: Integrated Research Application System)
Record Dates: First submitted 2016-01-20; First posted 2016-01-29 (Estimated); Results first posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-07

CONDITIONS: Widespread Chronic Pain
Keywords: Prevention trial; Cognitive Behaviour Therapy; CWP; Chronic widespread pain; RCT; Fibromyalgia; Prevention
MeSH Terms: conditions — Chronic Pain; Fibromyalgia | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Behavioural Therapy (Experimental): Brief Cognitive Behavioural Therapy delivered by telephone
  Interventions: Behavioral: Cognitive Behavioural Therapy
- Treatment as usual (No Intervention): The group allocated to usual care will receive no additional intervention - this will reflect the fact there is no specific intervention provided to patients currently for the prevention of CWP. Participants in this group will receive usual care and there will be no restriction on what this can involve. CBT is not readily available within the NHS and is generally restricted to persons who have developed specific conditions rather than persons at risk of those conditions.

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy — The CBT intervention, delivered by telephone, will consist of an initial assessment, 6 weekly sessions, and then booster sessions at 3 and 6 months. The intervention will be delivered by trained and accredited therapists. Participants will be supported by a self-management CBT manual. There will be a patient-centred assessment by the therapist for problem identification, risk assessment and development of a shared formulation of the current health problem. The sessions will involve education about musculoskeletal pain, somatic symptoms and specific CBT techniques such as pacing of activity, behavioural activation, diary keeping, identifying and challenging negative and unhelpful thinking patterns and the development of a longer term management plan.
  Other Names: Telephone-delivered Cognitive Behavioural Therapy
  Arms: Cognitive Behavioural Therapy

SUMMARY:
It is known from many studies that when patients have developed chronic widespread pain (CWP) or fibromyalgia that managing such symptoms is extremely challenging for both doctors and patients. The investigators have shown in a recently completed study funded by Arthritis Research UK that a course of Cognitive Behaviour Therapy delivered by telephone (tCBT) or an exercise regime can substantially improve the chances of the symptoms improving. The investigators now plan to offer this therapy to patients who are at a high risk of developing CWP (but who have not developed it yet) to see whether its onset can be prevented.

DETAILED DESCRIPTION:
Chronic widespread pain (CWP), the cardinal feature of fibromyalgia, is associated with lost work productivity, psychological ill health, and poor quality of life. It is one of the most common reasons for referral to a rheumatologist. The cost of CWP is high in terms of both individual, societal and health costs: for example, in the United States, mean per-patient costs (including pain and non-pain-related medication, physician consultations, tests and procedures, and emergency department visits) in the 6 months following a new diagnosis of fibromyalgia have been reported as $3481, comparable to patients with rheumatoid arthritis but resulting in worse quality of life. Current guidelines recommend pharmacological, physical, and psychological therapies although the importance attributed to individual therapies is inconsistent. There is good evidence for musculoskeletal pain conditions generally that the longer the duration of symptoms, the less likely that symptoms are to improve, including with specific interventions. This is particularly so for CWP which, once developed, is challenging to manage and effect improvement.

A systematic review and meta-analysis of randomised controlled trials (RCT) of Cognitive Behaviour Therapy (CBT) for patients with fibromyalgia concluded that CBT improves coping with pain, reduces depressed mood and healthcare-seeking behaviour in such patients. The delivery of CBT by telephone has been shown to be effective, acceptable and accessible. The MUSICIAN study, which the investigators have recently concluded, tested telephone delivered CBT (tCBT) and/or exercise for patients with chronic widespread pain consulting to their GP. Three months after the end of therapy, both interventions resulted in significantly better primary outcome measures (patient global health) than treatment as usual, but there was no significant additional benefit of receiving both interventions. Recent analyses have demonstrated these benefits are maintained 2 years after the end of therapy. The investigators have conducted a comprehensive literature review with the aim of identifying randomised trials which had the aim of preventing the onset either of CWP or fibromyalgia. This review did not identify any such published trials. Further, a search of 11 international clinical trials registers/databases (including US, UK, Europe, Australia/New Zealand, Japan), undertaken in Autumn 2013 did not identify any ongoing trial with the aim of preventing the onset of CWP (or fibromyalgia).

There are several reasons why it may be desirable to try to prevent CWP onset, namely that the majority of CWP patients do not have important symptom improvement with current management (even within trials). Prediction models from epidemiological studies have been developed to identify "high risk" patients, which makes such an approach feasible. Research using the General Practice Research Database has demonstrated that prior to receiving a diagnosis of fibromyalgia in primary care, persons have a long-term prior history of consultation with symptoms. Although this will be the first prevention trial in this area, the concept of prevention using CBT has been addressed in musculoskeletal disorders with respect to intervention in neck pain and low back pain before people become patients and in mental disorders.

The investigators have conducted prospective epidemiological studies which have demonstrated that it is possible to identify "high risk" groups. In the first study, a high risk group for CWP onset was identified on the basis of two factors: somatic awareness (using the Somatic Symptom Scale) and illness behaviour (using the Illness Behaviour Score). This was replicated in a second study conducted by the applicants. These "aetiological models" excluded pain and therefore the investigators have re-analysed data from the latter study (also considering pain status) to identify the best predictors of onset and which results in a model more suitable for use in prevention studies. The resulting "at risk model" requires regional pain and two of the following: maladaptive behavioural response to illness), a high number of somatic symptoms, and sleep disturbance. In the second "validation" study, from a population of 2,374 persons without CWP, 653 satisfied the definition of "high risk of CWP" of whom 139 had developed CWP twelve months later (that is a Positive Predictive value of 21.3%). Amongst persons not deemed to be at high risk (n=1721), 77 developed CWP which is a Negative Predictive Value of 95.5%.

The investigators have previously shown short and long-term effectiveness of tCBT for CWP (compared to usual care). Specifically this demonstrated sustained improvement in patient global assessment of change, reduced psychological distress, fear of movement and reliance on passive coping styles. Secondly the investigators have developed and refined statistical models which identify persons at high risk for the future development of CWP. The investigators therefore now propose a study to test whether tCBT can reduce the risk of CWP onset amongst those at high risk.

Three health boards in Scotland will be research sites for the study. The three health boards are NHS Grampian, NHS Highland, and NHS Greater Glasgow and Clyde. The study will require the involvement of 7 or 8 equivalent general practices. The investigators will mail a randomly selected sample of adults aged 25 years and over registered with participating general practices in the study areas. The Scottish Primary Care Research Network (SPCRN) will be involved in recruitment of patients to this study from primary care. SPCRN staff provide GP practices with an expert service to undertake searches of their electronic databases to identify a random sample of potentially eligible patients and prepare the ethically approved letters to be sent out. Searches are undertaken at each GP practice before the screening survey questionnaires are sent out by Health Informatics Centre Services in Dundee on behalf of the practice. Patients will return completed survey questionnaires to the research team at the University of Aberdeen where responses will be assessed by the research team for eligibility and patients sent invitation letters if eligible.

The "screening questionnaire" will determine whether a) respondents meet the study eligibility criteria and b) respondents would be willing to be contacted again regarding a treatment trial for "musculoskeletal health". The questionnaire will include:

* Pain assessed by specific questions on the experience of pain, consultation and body manikins (which will provide site and also allow us to exclude those who already have chronic widespread pain).
* Illness Behaviour Scale
* Somatic Symptoms Scale (excluding pain items)
* Sleep Problem Scale
* Quality of Life and Wellbeing
* General Health Questionnaire
* Chalder Fatigue Scale A list of eligible patients will be provided to the general practitioner in advance, with the option of indicating any as unsuitable for the study. Patients would then be sent information about the study and subsequently contacted by a member of the research team by telephone and, if appropriate, consented and recruited into the trial.

Included in the mailing to eligible patients will be an information sheet, consent form, and a best-time-to-call slip. Once a patient has returned a signed consent form and best-time-to-call slip, a member of the research team will phone them. The researcher will read out from a script giving information about the study, and the patient will have the opportunity then to ask questions about the study. If the patient consents to participate the participant will be recruited to the study and randomised to one of the arms of the trial.

Follow-up questionnaires will be mailed to participants at 3, 12 and 24 months after the treatment start date (for participants in the active treatment group) or dummy treatment start date (for those in usual care). Instruments included in the follow-up questionnaires will be the same as in the screening survey questionnaire. Additionally, follow-up questionnaires will include the Patient Global Impression of Change, and questions on health care usage.

Participants will have the option to withdraw from the treatment or the study at any time. Those withdrawing from the treatment will continue to be sent follow-up questionnaires unless the participant requests not to receive them. Failure of any participant to complete a follow-up questionnaire at any particular timepoint will not be counted as a withdrawal unless the participant requests not to receive any further follow-ups.

Our previous longitudinal study of onset of CWP (and subsequent replication) has suggested that 21% of "high risk" persons identified will develop CWP over the course of the next twelve months. Our previous data is based on persons with pain and at least 2 out of 3 other "risk factors". There are no published studies of prevention of CWP on which to base our measure of effect. However in the MUSICIAN study some subjects, although reporting CWP at the screening survey, no longer had CWP at the enrolment interview. These participants were however still eligible to take part, provided the participant had regional pain. Therefore those subjects with regional pain provide a sub-population on which to base the likely effects of the tCBT. Amongst such subjects, those who received tCBT had a reduced odds of having CWP at the end of the study OR 0.5 95% CI (0.2-1.4) compared to those in usual care.

Thus the study is powered on the ability of the current study to reduce the onset of CWP from 21% to 12%, with 90% power and a 5% significance level. The investigators further assume, based on prior data, that 75% of persons allocated to the tCBT arm will be adherent to the intervention, and that 80% of all subjects will return the follow-up questionnaires to assess outcome.

Accordingly the investigators require 473 subjects per arm that is a total of 946 subjects recruited. In MUSICIAN exactly 50% of those found eligible and willing to consider taking part ultimately were randomised. A previous trial of a cognitive-behavioural intervention to prevent chronic pain found that 36% of patients identified as eligible ended up being recruited to the study. If 80% of eligible patients agreed to be contacted about taking part, this equates to 45% of those eligible and willing to consider taking part being randomised - higher numbers for a clinical trial of CWP reflect the fact that this is a prevention trial rather than a treatment trial and may be less attractive to potential participants. Thus the investigators aim to find a total of 2102 subjects who are eligible and willing to consider taking part. Assuming a participation rate to the survey of 30%, that 1 in 4 people will be "at risk", and (using data from MUSICIAN) that 80% of people who return a questionnaire agree to consider taking part, the investigators require to survey 35 037 persons.

A pre-defined statistical analysis plan will be developed and signed off by the trial steering committee before undertaking any data analysis. Comparison between arms will be on an intention-to-treat basis (main analysis) with a per protocol sensitivity analysis.

Characteristics of the study participants in the two treatment arms will be described using simple summary statistics. Descriptive statistics will include mean and standard deviation for normally distributed continuous data, median and inter-quartile range for skewed continuous data and count and percentage for categorical data. No formal statistical comparisons will be made between baseline characteristics. Primary and secondary outcomes will be described at the three follow-up times: 3, 12 and 24 months, using appropriate summary statistics.

ELIGIBILITY:
Inclusion Criteria:

* A 'high-risk' profile for developing CWP as identified on the screening survey, i.e.:

  * Have pain for which the patient has sought consultation to primary care in the last 6 months
  * Any 2 of the following: Illness Behaviour Score > 4; Somatic Symptom Score > 2; Sleep Problem Score > 4
* Access to a land-line telephone or mobile telephone
* Ability to understand English sufficiently to participate in the intervention
* Ability to give informed consent
* Aged 25 years or over

Exclusion Criteria:

* Meeting American College of Rheumatology definition of CWP in the 1990 criteria for fibromyalgia (as assessed by the screening questionnaire)
* Medical conditions which would make the proposed intervention unsuitable (e.g. cognitive ability)

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1002 (Actual)
Dates: Start 2016-05; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary J Macfarlane, MBChB PhD MD, Principal Investigator — University of Aberdeen
Locations (3):
- United Kingdom (3):
  - NHS Grampian, Aberdeen
  - NHS Greater Glasgow & Clyde, Glasgow
  - NHS Highland, Inverness

IPD SHARING:
Plan to Share IPD: No
After completion of the study individual participant data will be made available to other researchers on request as decided by the study data management committee.

REFERENCES:
- [Derived] Macfarlane GJ, Beasley M, Scott N, Chong H, McNamee P, McBeth J, Basu N, Hannaford PC, Jones GT, Keeley P, Prescott GJ, Lovell K. Maintaining musculoskeletal health using a behavioural therapy approach: a population-based randomised controlled trial (the MAmMOTH Study). Ann Rheum Dis. 2021 Jul;80(7):903-911. doi: 10.1136/annrheumdis-2020-219091. Epub 2021 Feb 1. PMID 33526434
- [Derived] Fraser C, Beasley M, Macfarlane G, Lovell K. Telephone cognitive behavioural therapy to prevent the development of chronic widespread pain: a qualitative study of patient perspectives and treatment acceptability. BMC Musculoskelet Disord. 2019 May 10;20(1):198. doi: 10.1186/s12891-019-2584-2. PMID 31077168
- [Derived] Macfarlane GJ, Beasley M, Prescott G, McNamee P, Keeley P, Artus M, McBeth J, Hannaford P, Jones GT, Basu N, Norrie J, Lovell K. The Maintaining Musculoskeletal Health (MAmMOTH) Study: Protocol for a randomised trial of cognitive behavioural therapy versus usual care for the prevention of chronic widespread pain. BMC Musculoskelet Disord. 2016 Apr 26;17:179. doi: 10.1186/s12891-016-1037-4. PMID 27113442

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cognitive Behavioural Therapy | Treatment as Usual
Started | 501 | 501
Completed | 500 | 496
Not Completed | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Behavioural Therapy | Treatment as Usual | Total
Number analyzed (Participants) | 501 | 501 | 1002
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: There was 1 post-randomisation exclusion in the Cognitive Behavioural Therapy group and 5 post-randomisation exclusions in the Treatment as usual group.
  years
    number analyzed (Participants) | 500 | 496 | 996
    (all) | 58.8 [47.7 to 68.7] | 59.5 [47.9 to 68.9] | 59.3 [47.9 to 68.8]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: There was 1 post-randomisation exclusion in the Cognitive Behavioural Therapy group and 5 post-randomisation exclusions in the Treatment as usual group.
  Participants
    number analyzed (Participants) | 500 | 496 | 996
    Female | 209 | 204 | 413
    Male | 291 | 292 | 583
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Development of Chronic Widespread Pain Assessed by Questionnaire
Description: The development of new chronic widespread pain, as defined by ACR 1990 criteria for fibromyalgia and assessed by questionnaire, at follow-up will be compared between participants in the two treatment arms. A participant was counted as having chronic widespread pain if they said they had pain in the last month that had lasted a day or more, indicated on a paper manikin that the pain that was on both the left and right hand sides, and above and below the waist, and in the axial skeleton, and answered that they had this pain for more than 3 months. If they did not have pain that was that above and below the waist and on the left and right hand sides, and in the axial skeleton, or they did not say they had the pain for more than 3 months, then they did not have chronic widespread pain.
Time Frame: 12 months after treatment start
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitive Behavioural Therapy | Treatment as Usual
Number analyzed (Participants) | 384 | 441
Participants | 69 | 77

2. Secondary Outcome: Pain Assessed by Questionnaire
Description: Assessed by follow-up questionnaire. Participants were asked if they had pain in the last month that had lasted a day or more and could answer 'yes' or 'no.
Time Frame: 3 months after treatment start
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitive Behavioural Therapy | Treatment as Usual
Number analyzed (Participants) | 380 | 443
Participants | 308 | 384

3. Secondary Outcome: Pain Assessed by Questionnaire
Description: Assessed by follow-up questionnaire. Participants were asked if they had pain in the last month that lasted a day or more, and could answer 'yes' or 'no'.
Time Frame: 12 months after treatment start
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitive Behavioural Therapy | Treatment as Usual
Number analyzed (Participants) | 384 | 441
Participants | 305 | 373

4. Secondary Outcome: Pain Assessed by Questionnaire
Description: as for outcome 3
Time Frame: 24 months after treatment start
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitive Behavioural Therapy | Treatment as Usual
Number analyzed (Participants) | 400 | 453
Participants | 305 | 376

5. Secondary Outcome: Illness Behaviour Assessed by Illness Behaviour Scale
Description: Illness Behaviour Scale, which is comprised of the 'Treatment experiences' and 'Effects of symptoms' sub-scales of the Illness Attitudes Scales. The range of scores is from 0 (best) to 24 (worst).
Time Frame: 3 months after treatment start
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Behavioural Therapy | Treatment as Usual
Number analyzed (Participants) | 379 | 441
score on a scale | 8.96 (3.99) | 9.21 (3.86)

6. Secondary Outcome: Illness Behaviour Assessed by Illness Behaviour Scale
Description: as for outcome 5
Time Frame: 12 months after treatment start
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Behavioural Therapy | Treatment as Usual
Number analyzed (Participants) | 373 | 431
score on a scale | 8.21 (4.04) | 8.96 (4.19)

7. Secondary Outcome: Illness Behaviour Assessed by Illness Behaviour Scale
Description: as for outcome 5
Time Frame: 24 months after treatment start
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Behavioural Therapy | Treatment as Usual
Number analyzed (Participants) | 310 | 377
score on a scale | 7.75 (4.14) | 8.95 (4.18)

8. Secondary Outcome: Somatic Symptom Reporting Assessed by Somatic Symptoms Scale
Description: Somatic Symptoms Scale, which measures the presence or absence of 5 somatic symptoms, with a range of 0 (best) to 5 (worst) somatic symptoms.
Time Frame: 3 months after treatment start
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitive Behavioural Therapy | Treatment as Usual
Number analyzed (Participants) | 379 | 442
Participants
  0 | 224 | 239
  1 | 96 | 127
  2-5 | 59 | 76

9. Secondary Outcome: Somatic Symptom Reporting Assessed by Somatic Symptoms Scale
Description: as for outcome 8
Time Frame: 12 months after treatment start
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitive Behavioural Therapy | Treatment as Usual
Number analyzed (Participants) | 372 | 432
Participants
  0 | 210 | 228
  1 | 103 | 123
  2-5 | 59 | 81

10. Secondary Outcome: Somatic Symptom Reporting Assessed by Somatic Symptoms Scale
Description: as for outcome 8
Time Frame: 24 months after treatment start
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitive Behavioural Therapy | Treatment as Usual
Number analyzed (Participants) | 310 | 377
Participants
  0 | 184 | 219
  1 | 82 | 90
  2-5 | 44 | 68

11. Secondary Outcome: Sleep Problems Assessed by Sleep Problem Scale
Description: Sleep Problem Scale
Time Frame: 3 months after treatment start
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Behavioural Therapy | Treatment as Usual
Number analyzed (Participants) | 377 | 439
score on a scale | 8.54 (4.99) | 9.16 (5.08)

12. Secondary Outcome: Sleep Problems Assessed by Sleep Problem Scale
Description: Sleep Problem Scale, with a range of 0 (best) to 20 (worst).
Time Frame: 12 months after treatment start
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Behavioural Therapy | Treatment as Usual
Number analyzed (Participants) | 373 | 432
score on a scale | 8.20 (4.89) | 9.20 (5.16)

13. Secondary Outcome: Sleep Problems Assessed by Sleep Problem Scale
Description: Sleep Problem Scale, with a range of 0 (best) to 20 (worst).
Time Frame: 24 months after treatment start
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Behavioural Therapy | Treatment as Usual
Number analyzed (Participants) | 309 | 376
score on a scale | 8.45 (5.3) | 9.06 (5.0)

14. Secondary Outcome: EQ-5D
Description: The EQ-5D is a standardised measure of health-related quality of life, with a range of values from 0 (worst) to 1 (best).
Time Frame: 3 months after treatment start
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Cognitive Behavioural Therapy | Treatment as Usual
Number analyzed (Participants) | 379 | 442
score on a scale | 0.74 [0.67 to 0.84] | 0.74 [0.65 to 0.84]

15. Secondary Outcome: EQ-5D
Description: as for outcome 14
Time Frame: 12 months after treatment start
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Cognitive Behavioural Therapy | Treatment as Usual
Number analyzed (Participants) | 371 | 435
score on a scale | 0.74 [0.66 to 0.84] | 0.74 [0.65 to 0.82]

16. Secondary Outcome: EQ-5D
Description: as for outcome 14
Time Frame: 24 months after treatment start
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Cognitive Behavioural Therapy | Treatment as Usual
Number analyzed (Participants) | 313 | 386
score on a scale | 0.74 [0.68 to 0.84] | 0.74 [0.65 to 0.84]

17. Secondary Outcome: Wellbeing
Description: ICECAP-A (ICEpop CAPability measure for Adults) is a self-report measure of capability wellbeing for adults, with a range of scores from -0.001 (worst) to 1 (best).
Time Frame: 3 months after treatment start
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Cognitive Behavioural Therapy | Treatment as Usual
Number analyzed (Participants) | 378 | 440
score on a scale | 0.89 [0.80 to 0.95] | 0.89 [0.78 to 0.95]

18. Secondary Outcome: Wellbeing
Description: as for outcome 17
Time Frame: 12 months after treatment start
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Cognitive Behavioural Therapy | Treatment as Usual
Number analyzed (Participants) | 368 | 429
score on a scale | 0.91 [0.82 to 0.97] | 0.89 [0.78 to 0.95]

19. Secondary Outcome: Wellbeing
Description: as for outcome 17
Time Frame: 24 months after treatment start
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Cognitive Behavioural Therapy | Treatment as Usual
Number analyzed (Participants) | 311 | 386
score on a scale | 0.91 [0.80 to 0.96] | 0.89 [0.79 to 0.95]

20. Secondary Outcome: Psychological Distress Assessed by GHQ-12
Description: GHQ-12 (12-item General Health Questionnaire) has a range of 0 (best) to 12 (worst).
Time Frame: 3 months after treatment start
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitive Behavioural Therapy | Treatment as Usual
Number analyzed (Participants) | 374 | 439
Participants
  0 | 224 | 207
  1 | 50 | 63
  2-5 | 65 | 96
  6-12 | 35 | 73

21. Secondary Outcome: Psychological Distress Assessed by GHQ-12
Description: GHQ-12 (12-item General Health Questionnaire) has a range of 0 (best) to 12 (worst).
Time Frame: 12 months after treatment start
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitive Behavioural Therapy | Treatment as Usual
Number analyzed (Participants) | 369 | 432
Participants
  0 | 201 | 202
  1 | 59 | 54
  2-5 | 68 | 113
  6-12 | 41 | 63

22. Secondary Outcome: Psychological Distress Assessed by GHQ-12
Description: GHQ-12 (12-item General Health Questionnaire) has a range of 0 (best) to 12 (worst).
Time Frame: 24 months after treatment start
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitive Behavioural Therapy | Treatment as Usual
Number analyzed (Participants) | 310 | 376
Participants
  0 | 168 | 178
  1 | 36 | 42
  2-5 | 67 | 91
  6-12 | 39 | 65

23. Secondary Outcome: Patient Global Impression of Change Assessed by 7-item Scale
Description: 7-item scale from "very much worse" to "very much better"
Time Frame: 3 months after treatment start
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitive Behavioural Therapy | Treatment as Usual
Number analyzed (Participants) | 378 | 442
Participants
  Very much better | 14 | 15
  Much better | 76 | 48
  A little better | 132 | 91
  No change | 100 | 165
  A little worse | 45 | 98
  Much worse | 11 | 23
  Very much worse | 0 | 2

24. Secondary Outcome: Patient Global Impression of Change Assessed by 7-item Scale
Description: 7-item scale from "very much worse" to "very much better"
Time Frame: 12 months after treatment start
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitive Behavioural Therapy | Treatment as Usual
Number analyzed (Participants) | 371 | 429
Participants
  Very much better | 24 | 15
  Much better | 88 | 59
  A little better | 90 | 84
  No change | 83 | 126
  A little worse | 65 | 119
  Much worse | 18 | 23
  Very much worse | 3 | 3

25. Secondary Outcome: Patient Global Impression of Change Assessed by 7-item Scale
Description: 7-item scale from "very much worse" to "very much better"
Time Frame: 24 months after treatment start
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitive Behavioural Therapy | Treatment as Usual
Number analyzed (Participants) | 378 | 442
Participants
  Very much better | 14 | 15
  Much better | 76 | 48
  A little better | 132 | 91
  No change | 100 | 165
  A little worse | 45 | 98
  Much worse | 11 | 23
  Very much worse | 0 | 2

26. Secondary Outcome: Fatigue Assessed by Chalder Fatigue Scale
Description: Chalder Fatigue Scale has a range of 0 (best) to 33 (worst).
Time Frame: 3 months after treatment start
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Behavioural Therapy | Treatment as Usual
Number analyzed (Participants) | 372 | 440
score on a scale | 12.2 (4.2) | 13.6 (4.2)

27. Secondary Outcome: Fatigue Assessed by Chalder Fatigue Scale
Description: Chalder Fatigue Scale has a range of 0 (best) to 33 (worst).
Time Frame: 12 months after treatment start
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Behavioural Therapy | Treatment as Usual
Number analyzed (Participants) | 370 | 433
score on a scale | 12.6 (4.5) | 13.6 (4.4)

28. Secondary Outcome: Fatigue Assessed by Chalder Fatigue Scale
Description: Chalder Fatigue Scale has a range of 0 (best) to 33 (worst).
Time Frame: 24 months after treatment start
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Behavioural Therapy | Treatment as Usual
Number analyzed (Participants) | 309 | 377
score on a scale | 13.0 (4.3) | 13.9 (4.4)

29. Secondary Outcome: Health Care Usage Assessed by Questionnaire
Description: Health care usage will be assessed by questionnaire at 3 months, 12 months and 24 months after treatment start to determine the cost-effectiveness of the intervention. Only the cost of health care usage for the 24 month period after treatment start was calculated using this data.
Time Frame: 24 months after treatment start
Measure: Mean (95% Confidence Interval); unit: £
Arm/Group | Cognitive Behavioural Therapy | Treatment as Usual
Number analyzed (Participants) | 277 | 343
£ | 3094.68 [1775.65 to 9074.15] | 3052.38 [1735.77 to 8567.24]

30. Secondary Outcome: Development of Chronic Widespread Pain Assessed by Questionnaire
Description: as for outcome 1
Time Frame: 3 months after treatment start
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitive Behavioural Therapy | Treatment as Usual
Number analyzed (Participants) | 380 | 443
Participants | 68 | 75

31. Secondary Outcome: Development of Chronic Widespread Pain Assessed by Questionnaire
Description: as for outcome 1
Time Frame: 24 months after treatment start
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitive Behavioural Therapy | Treatment as Usual
Number analyzed (Participants) | 400 | 453
Participants | 78 | 101

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Cognitive Behavioural Therapy | Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 3/501 | 9/501
Serious Adverse Events (participants affected / at risk) | 0/501 | 0/501
Other Adverse Events (participants affected / at risk) | 3/501 | 0/501
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cognitive Behavioural Therapy (N=501) | Treatment as Usual (N=501)
Participant expressing thoughts that might be considered suicidal to therapist or on questionnaire (Psychiatric disorders) | 2 | NA
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-05-22): https://cdn.clinicaltrials.gov/large-docs/03/NCT02668003/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-19): https://cdn.clinicaltrials.gov/large-docs/03/NCT02668003/SAP_001.pdf